CLINICAL TRIAL: NCT02176590
Title: Improving Family Well-Being and Child School Readiness: Power PATH Dual Generation Intervention With Head Start Preschoolers and Their Parents
Brief Title: Improving Family Well-Being and Child School Readiness: Power PATH Dual Generation Intervention
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90YR0075
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Power PATH; Head Start as Usual
Keywords: PATHS Social Emotional Learning; Coping Power; Power PATH; Head Start
MeSH Terms: interventions — Schools, Nursery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Power PATH (Experimental): Classroom PATHS Social Emotional Learning Curriculum (for preschool classrooms) plus Coping Power parent intervention (teaches parents what children are learning in the classroom PATHS program and also provides parents with mental health intervention and parenting topics to promote family well-being)
  Interventions: Behavioral: Power PATH
- Head Start as usual (Active Comparator): Head Start as usual (will measure the effects of Head Start programming as usual on the primary outcomes)
  Interventions: Other: Head Start as usual

INTERVENTIONS:
Behavioral: Power PATH — PATHS: Teacher-led classroom curriculum promoting a positive classroom environment and teaching social-emotional skills
  Other Names: Promoting Alternative Thinking Strategies (PATHS) Preschool/Kindergarten Social Emotional Learning Classroom Curriculum; Coping Power parent program
  Arms: Power PATH
Other: Head Start as usual — Standard Head Start programming (including classroom instruction, meals, and family services)
  Arms: Head Start as usual

SUMMARY:
This project will test the proximal and distal effects of an integrated dual-generation intervention, Power PATH, in Head Start preschoolers and their parents in Alabama.

DETAILED DESCRIPTION:
This project will test the proximal and distal effects of an integrated dual-generation intervention approach, Power PATH, in an existing Head Start University Partnership in Alabama. Dual generation approaches recognize the need to intervene with both parents and children in Head Start preschools, in order to improve parents' ability to provide safe and supportive caregiving environments and to prepare children for the transition to elementary school academically and behaviorally. Parents of Head Start preschoolers often have high levels of poverty, stress, and mental health needs (Yoshikowa, Aber, & Beardslee, 2012) and their children are at-risk for academic, behavioral, and social-emotional difficulties (Aber, Jones, & Cohen, 2000; Costello, Keeler, & Angold, 2001; Morales & Guerra, 2006). Thus, in this project, two evidence-based and widely-utilized preventive interventions will be adapted and thoughtfully integrated, in collabo-ration with Head Start personnel, to provide intensive, high quality services to Head Start parents and children. First, the Power PATH Parent Intervention program, adapted from Coping Power (Wells, Lochman & Lenhart, 2008) for this dual-generation approach, will be implemented to address parental mental health needs, to increase parental employment and financial security, and to improve parents' ability to model effective social-emotional skills. The parent intervention will help parents create a positive and predictable home environment, and support their child's academic learning and emotional and behavioral self-regulation. Second, the Promoting Alterna-tive Thinking Strategies (PATHS) Preschool Social and Emotional Learning curriculum (Domitrovich et al., 1999) will be implemented in the preschool classrooms. PATHS is a universal, classroom-based curriculum that increases children's social-emotional competence and self-regulatory skills, leading to long-term social, behavioral and academic gains. The Power PATH program will incorporate both of these parent and child interventions, and will include opportuni-ties for the children to teach their parents the social and emotional skills they are learning in the classroom, to promote skill- generalization and transfer to the home environment. This study will also identify novel intervention mediators and moderators, essential for interrupting the intergen-erational transmission of chronic social stress, and will identify the best interventions for families, particularly during preschool when self-regulation skills are still malleable, and children's primary environments and physiological responses to stress are likely to moderate intervention effects (Bierman et al., 2008; Boyce & Ellis, 2005; Porges, 2007). In summary, addressing sources of chronic stress in the parents of Head Start preschoolers (i.e., employment and financial insecurity, mental health needs, and family stressors) through the Power PATH dual generation intervention is expected to prepare parents to better support, shape and model their children's self-regulation skills and to better foster their children's school readiness, and to improve overall family well-being.

ELIGIBILITY:
Inclusion Criteria:

* 4 year old preschool students in participating Head Start centers/classrooms in West Central Alabama, and their parents and teachers

Exclusion Criteria:

* Severe developmental delay (making the student unable to complete the primary study measures)

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 540 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Child School Readiness | One year (repeated through 1st grade)
  Indicators of child school readiness (Behavior, Executive Functioning, Emotional Regulation, Pre-Reading skills) will be assessed at the end of preschool.
Family Well-being | One Year (repeated through 1st grade)
  Indicators of Family Well-Being will be measured at the end of preschool (Parental stress, parenting, parental depression, economic and financial security, family environment)

CONTACTS AND LOCATIONS:
Overall Officials: Ansley Gilpin, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Tuscaloosa, Alabama, United States